CLINICAL TRIAL: NCT02123147
Title: Examining the Immunological Process of Autoimmune Patients
Status: Withdrawn | Type: Observational
Why Stopped: due to the lack of funding to continue
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400079
Record Dates: First submitted 2014-04-16; First posted 2014-04-25 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Sjogren's Syndrome; Autoimmune Diseases; Dry Eyes; Dry Mouth
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases; Dry Eye Syndromes; Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sjogren's syndrome: Patients who are diagnosed with Sjogren's syndrome. Blood will be collected once every 3-6 months for up to 3 years.
- Healthy Control: Patients who are diagnosed with healthy control. Blood will be collected once every 6 months for up to 3 years.

SUMMARY:
Sjögren's syndrome (SjS) is an autoimmune disease characterized primarily by exocrine gland dysfunction, specifically of the salivary and lacrimal glands, resulting in dry mouth and dry eyes symptoms. It can be systemic by affecting other organs including the gastrointestinal tract, skin, lungs, vasculature, kidneys, bladder and vagina. Involvement of the musculature can lead to fibromyalgia-like symptoms and chronic fatigue, while approximately 20% of patients develop various neuropathies, including sensory, peripheral, cranial and myelopathic neuropathies exhibited by cognitive impairments such as dementia, lack of concentration, memory loss and various psychiatric disorders. Like most autoimmune connective tissue diseases, SjS shows a sexual dimorphism with women affected 10-times more frequently than men, suggesting a role for sex hormones in disease susceptibility or progression. One common feature of SjS is it infiltration of mononuclear cells into the salivary and lacrimal glands, aggregating into clusters referred to as lymphocytic foci (LF). Critical to the studies proposed is the fact that a predominant cell population of LF is the pathogenic TH17 cell that produces IL-17 cytokine and autoreactive B cells reactive to M3R, Ro, and La autoantigens. The goal of this study is characterize the change in receptor gene repertoires of autoreactive B and T cells at different time points during the disease process and examine the correlation with various disease parameters.

DETAILED DESCRIPTION:
Blood from patient and healthy controls will be collected once every 3-6 months. White blood cells from blood samples will be separated. Tests will be done to see which substances these cells make. Using sequencing techniques, the investigators will determine the genetic code of the receptors expressed on these cells. The investigators plan to test how these cells change over the period of at least 3 years at different visits. In addition, the investigators will check how these changes relate to patients' general medical history relevant to autoimmune disease, lab results and physical examinations and exams pertinent to the diagnosis of autoimmune disease, and psychosocial data.

ELIGIBILITY:
Inclusion Criteria for Sjogren's syndrome patients:

* Primary Sjogren's syndrome patients: primary Sjogren's syndrome patients who meet the revised criteria for SjS diagnosis by the American-European Consensus Group.
* Secondary Sjogren's syndrome patients: secondary Sjogren's syndrome patients who meet the criteria for primary Sjogren's syndrome in association with other autoimmune diseases such as systemic lupus erythematosus , dermatomyositis, scleroderma, idiopathic arthritis, mixed connective tissue disease, etc.

Inclusion Criteria for healthy controls:

-Subjects who does not have history of autoimmune diseases.

Exclusion Criteria:

* Pregnant women.
* Patients with history of lymphoma or malignancy.

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 150 Sjogren's syndrome patients and 50 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Receptor gene rearrangement. | Every 3 months for 3 years
  Gene arrangement of the receptors in patients will be assessed every 3 months for 3 years.
Receptor gene rearrangement | Every 6 months for 3 years.
  Gene arrangement of the receptors in healthy controls will be assessed every 6 months for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Cuong Nguyen, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States